CLINICAL TRIAL: NCT03147079
Title: Mighty Mums - a Lifestyle Intervention at Primary Care Level for Pregnant Women With Obesity
Brief Title: Study of Antenatal Care Intervention Directed to Pregnant Women With Obesity
Acronym: Mighty Mums
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FoU-project id 203431; 505-10 (Other: Approval number from the ethical review board)
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Obesity Complicating Childbirth
Keywords: obesity; pregnancy; lifestyle; gestational weight gain; weight of offspring; antenatal care; health behavior; physical activity; diet; programme evaluation; costs and costs analysis
MeSH Terms: conditions — Obesity; Gestational Weight Gain; Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Open intervention study with 2 control arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Lifestyle intervention
  Interventions: Behavioral: Lifestyle intervention
- Internal controls (Experimental)
  Interventions: Behavioral: Lifestyle intervention
- External controls (Experimental)
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention

SUMMARY:
The purpose of this study is to determine whether a behavioural intervention focusing on diet and physical activity is cost-effective in decreasing weight gain during pregnancy among pregnant women with body mass index above 30, and has effect on the weight of offspring at birth and at 2.5 years of age

DETAILED DESCRIPTION:
Obesity in relation to pregnancy is becoming an increasing public health issue and 48% of women assigned to antenatal care in Sweden have overweight (BMI≥25) or obesity (BMI≥30). Obesity is associated with adverse perinatal outcomes, the risks increase with increasing BMI and excessive gestational weight gain (GWG) further increases the risks of adverse pregnancy outcomes. Lifestyle intervention can help pregnant women with obesity to limit their GWG. This study evaluated whether a low-budget antenatal lifestyle intervention programme, with emphasis on nutrition and physical activity, influenced GWG and maternal and perinatal outcomes for pregnant women with obesity. The study also evaluated which specific components of the intervention that had effect.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* BMI>30

Exclusion Criteria:

* first antenatal care visit after week 20 of the pregnancy
* abortion
* miscarriage

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1354 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain < 7 kg | 7 months
  Weight gain measured from enrollment/first antenatal care visit to last visit before partum, measured in kg

CONTACTS AND LOCATIONS:
Overall Officials: Marie Berg, RN PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska Academy, Institute of Health Care Sciences, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dencker A, Premberg A, Olander EK, McCourt C, Haby K, Dencker S, Glantz A, Berg M. Adopting a healthy lifestyle when pregnant and obese - an interview study three years after childbirth. BMC Pregnancy Childbirth. 2016 Jul 30;16(1):201. doi: 10.1186/s12884-016-0969-x. PMID 27473076
- [Background] Petrov Fieril K, Fagevik Olsen M, Glantz A, Larsson M. Experiences of exercise during pregnancy among women who perform regular resistance training: a qualitative study. Phys Ther. 2014 Aug;94(8):1135-43. doi: 10.2522/ptj.20120432. Epub 2014 May 1. PMID 24786941
- [Background] Haby K, Glantz A, Hanas R, Premberg A. Mighty Mums - An antenatal health care intervention can reduce gestational weight gain in women with obesity. Midwifery. 2015 Jul;31(7):685-92. doi: 10.1016/j.midw.2015.03.014. Epub 2015 Apr 9. PMID 25912510
- [Derived] Haby K, Gyllensten H, Hanas R, Berg M, Premberg A. A Lifestyle Intervention During Pregnancy and Its Effects on Child Weight 2.5 Years Later. Matern Child Health J. 2022 Sep;26(9):1881-1890. doi: 10.1007/s10995-022-03395-5. Epub 2022 Mar 6. PMID 35253077
- [Derived] Gyllensten H, Haby K, Berg M, Premberg A. Cost effectiveness of a controlled lifestyle intervention for pregnant women with obesity. BMC Pregnancy Childbirth. 2021 Sep 21;21(1):639. doi: 10.1186/s12884-021-04098-5. PMID 34548038
- [Derived] Haby K, Berg M, Gyllensten H, Hanas R, Premberg A. Mighty Mums - a lifestyle intervention at primary care level reduces gestational weight gain in women with obesity. BMC Obes. 2018 Jun 4;5:16. doi: 10.1186/s40608-018-0194-4. eCollection 2018. PMID 29881627